CLINICAL TRIAL: NCT04765657
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Inclisiran in Asian Patients With ASCVD or ASCVD High Risk and Elevated Low-density Lipoprotein Cholesterol as an Adjunct to Diet and Maximally Tolerated Statins With or Without Additional Lipid-lowering Therapy (ORION-18)
Brief Title: Study of Efficacy and Safety of Inclisiran in Asian Participants With Atherosclerotic Cardiovascular Disease (ASCVD) or ASCVD High Risk and Elevated Low Density Lipoprotein Cholesterol (LDL-C)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CKJX839A12307
Record Dates: First submitted 2021-02-05; First posted 2021-02-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hypercholesterolemia
Keywords: inclisiran; siRNA; dyslipidemia; KJX839
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inclisiran sodium 300 mg (Experimental): Subcutaneous injection
  Interventions: Drug: inclisiran sodium
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: inclisiran sodium — Subcutaneously injected on Day 1, 90 and 270 (Core Part). Subcutaneously injected on Day 360 and every 6 months thereafter until EOS visit (Extension Part)
  Other Names: KJX839
  Arms: inclisiran sodium 300 mg
Drug: Placebo — Subcutaneously injected on Day 1, 90, and 270.
  Arms: Placebo

SUMMARY:
A multicenter study to evaluate safety and efficacy of inclisiran in Asian patients with ASCVD or ASCVD high risk and elevated LDL-C

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate the efficacy and safety of inclisiran sodium 300mg to support the indication for LDL-C reduction of inclisiran in Asian patients with atherosclerotic cardiovascular disease (ASCVD) or ASCVD-high risk patients with elevated LDL-C as an adjunct to diet and maximally tolerated dose statins with or without additional lipid-lowering therapy.

A core part (2-week screening period and a 12-month double-blinded treatment period), and an extension part (until reasonable access to the IMP post product launch provided for the participants)

ELIGIBILITY:
Inclusion Criteria:

-At screening participants with: ASCVD (including acute coronary syndrome (ACS), stable coronary heart disease, post revascularization, ischemic cardiomyopathy, ischemic stroke, transient ischemic attack (TIA), and peripheral atherosclerosis) and Serum LDL-C ≥1.8 mmol/L (≥70 mg/dL) OR ASCVD high risk (LDL-C ≥4.9 mmol/L, diabetes, high 10-year ASCVD risk assessed by Chinese ASCVD Risk Assessment Flow Chart , or high risk per local guidelines with a target LDL-C of <100 mg/dL) and Serum LDL-C ≥2.6 mmol/L (≥100 mg/dL)

* Fasting triglyceride < 400 mg/dL (< 4.52 mmol/L) at screening.
* Participants on statins should be receiving a maximally tolerated dose . Maximum tolerated dose is defined as the maximum dose of statin that can be taken on a regular basis without intolerable AE. Intolerance to any dose of statin must be documented as historical AEs attributed to the statin in question on the source documentation and on the Medical history page of the eCRF
* Participants not receiving statin must have a documented evidence of intolerance to all doses of at least 2 different statins(or the corresponding local definition of complete intolerance to statins)
* Participants following lifestyle modification should be on the therapy of LDL-C lowering (such as statin monotherapy, or statin incombination with ezetimibe) with a stable dose for ≥30 days before screening and have no planned medication or dose change during study participation.
* Participants are willing and able to give informed consent before initiation of any study related procedures and willing to comply with all required study procedures.

Exclusion Criteria:

* New York Heart Association (NYHA) class IV heart failure or last known left ventricular ejection fraction <25%.
* Cardiac arrhythmia with clinical significance within 3 months prior to randomization that is not controlled by medication or via ablation.
* Major adverse cardiovascular event within 3 months prior to randomization.
* Uncontrolled severe hypertension: systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg prior to randomization despite antihypertensive therapy.
* Calculated glomerular filtration rate ≤30 mL/min by estimated glomerular filtration rate (eGFR) using standardized clinical methodology.
* Severe concomitant non-cardiovascular disease that carries the risk of reducing life expectancy to less than 2 years.
* History of malignancy that required surgery (excluding local and wide-local excision), radiation therapy and/or systemic therapy during the three years prior to randomization.
* Barrier method: Condom or Occlusive cap (e.g. diaphragm or cervical/vault caps).
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Core: Percentage change in low- density lipoprotein cholesterol (LDL-C) | Baseline, Day 330
  Superiority of inclisiran compared to placebo in reducing LDL-C from baseline to Day 330
Extension: Number of participants with Adverse Events | Day 360 until study completion, an average of 3 years
  Evaluation of the safety and tolerability of inclisiran, treatment emergent Adverse events and Serious Adverse Events

SECONDARY OUTCOMES:
Core: Time adjusted percentage change in LDL-C | From baseline after Day 90 and up to Day 360
  The superiority of inclisiran compared to placebo in reducing LDL-C from baseline to Day 330 and over time
Core: Absolute change in LDL-C | From baseline to Day 330
  The superiority of inclisiran compared to placebo in reducing LDL-C from baseline to Day 330 and over time
Core: Time adjusted absolute change in LDL-C | From baseline after Day 90 and up to Day 360
  The superiority of inclisiran compared to placebo in reducing LDL-C from baseline to Day 330 and over time
Core: Percentage change in PCSK9 | From baseline to Day 330
  The superiority of inclisiran compared to placebo in reducing PCSK9 from baseline to Day 330
Core: Absolute change in PCSK9 | From baseline to Day 330
  The superiority of inclisiran compared to placebo in reducing PCSK9 from baseline to Day 330
Core: Proportion of participants reaching LDL-C levels of <25 mg/dL, <50 mg/dL, <70 mg/dL, and <100 mg/dL | Day 330
  The superiority of inclisiran compared to placebo in individual response rate for lipid controlling
Core: Proportion of participants in each group with ≥ 50% LDL-C reduction | From baseline to Day 330
  The superiority of inclisiran compared to placebo in individual response rate for lipid controlling
Core: Proportion of participants in each group who attain global lipid targets for their level of ASCVD risk (55mg/dl for ASCVD patients, 70mg/dl for ASCVD high risk patients) | Day 330
  The superiority of inclisiran compared to placebo in individual response rate for lipid controlling
Core: Percentage change in total cholesterol, ApoB, non-HDL-C, ApoA1, HDL-C, Lp(a) and triglycerides | From baseline to Day 330
  The superiority of inclisiran compared to placebo in reducing other lipids, lipoproteins and apolipoproteins
Core: Absolute change in total cholesterol, ApoB, non-HDL-C, ApoA1, HDL-C, Lp(a) and triglycerides | From baseline to Day 330
  The superiority of inclisiran compared to placebo in reducing other lipids, lipoproteins and apolipoproteins

CONTACTS AND LOCATIONS:
Locations (31):
- China (21):
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Foshan, Guangdong
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Hohhot, Inner Mongolia
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nantong, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Xuzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Zhujing, Shanghai Municipality
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Xiamen
- Novartis Investigative Site, Singapore, Singapore
- South Korea (7):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Incheon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Seoul, South Korea
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Huo Y, Lesogor A, Lee CW, Chiang CE, Mena-Madrazo J, Poh KK, Jeong MH, Maheux P, Zhang M, Wei S, Han Y, Li Y. Efficacy and Safety of Inclisiran in Asian Patients: Results From ORION-18. JACC Asia. 2023 Nov 14;4(2):123-134. doi: 10.1016/j.jacasi.2023.09.006. eCollection 2024 Feb. PMID 38371290